CLINICAL TRIAL: NCT01065337
Title: Study on Induced Wound Healing Through Application of Expanded Autologous Bone Marrow Stem Cells in Diabetic Patients With Ischemia-induced Chronic Tissue Ulcers Affecting the Lower Limbs
Brief Title: Induced Wound Healing by Application of Expanded Bone Marrow Stem Cells in Diabetic Patients With Critical Limb Ischemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Diethelm Tschoepe, Prof. Dr. Dr., Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDZ-SBE-2004
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Diabetic Foot
Keywords: peripheral arterial occlusion disease (PAD); diabetic foot; critical limb ischemia (CLI); stem cell therapy
MeSH Terms: conditions — Diabetic Foot; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- control group (No Intervention): patients received standard of care wound treatment according guideline of the American Diabetes Association (ADA)
- bone marrow stem cells intraarterial (Active Comparator): bone marrow stem cells administered intraarterial
  Interventions: Biological: bone marrow stem cells (BMC)
- tissue repair cells intramuscular (Active Comparator): expanded bone marrow cells enriched in CD90+ mesenchymal stem cells administered intramuscular
  Interventions: Biological: tissue repair cells (TRC)
- tissue repair cells intraarterial (Active Comparator): expanded bone marrow cells enriched in CD90+ mesenchymal stem cells administered intraarterial
  Interventions: Biological: tissue repair cells (TRC)
- bone marrow stem cells intramuscular (Active Comparator): bone marrow stem cells administered intramuscular
  Interventions: Biological: bone marrow stem cells (BMC)

INTERVENTIONS:
Biological: tissue repair cells (TRC) — expanded bone marrow cells enriched in CD90+ mesenchymal stem cells
  Arms: tissue repair cells intraarterial; tissue repair cells intramuscular
Biological: bone marrow stem cells (BMC) — bone marrow stem cells
  Arms: bone marrow stem cells intraarterial; bone marrow stem cells intramuscular

SUMMARY:
Diabetic foot patients with chronic limb ischemia and without the option for surgical or interventional revascularization were recruited and randomized to the transplant groups or the control group within this clinical trial. These patients are randomized to control or intervention group, whereas the intervention is divided into bone marrow cells administered intramuscular or intraarterial or expanded bone marrow cells administered intramuscular or intraarterial resulting in five distinct groups. To measure the therapeutic effects of the various treatment arms patients were evaluated for (ankle brachial index (ABI), transcutaneous oxygen partial pressure (TcPO2), and reactive hyperemia (Blood Oxygen Level Dependent [BOLD]). Patients also underwent imaging with angiographic methods.

DETAILED DESCRIPTION:
Diabetic foot (DF) is a concomitant illness of diabetes mellitus. Diabetes is one of the main causes of non-traumatic amputation worldwide due to severe peripheral arterial occlusive disease with chronic critical limb ischemia being the most abundant problem. Ulceration occurs as failure of oxygenation, nutrient supply and progressive occlusion of larger blood vessels often exacerbates pre-existing microvascular abnormalities.

Purified bone marrow mononuclear cells or expanded bone marrow cells enriched in Cluster of Differentiation 90+ (CD90+) mesenchymal stem cells (named tissue repair cells, [TRCs]) are used in the treatment of diabetic ulcers in comparison to bone marrow derived stem cells to induce revascularization of the affected limb and to enhance local perfusion. Cells are administered intramuscular or intraarterial. A control group of patients treated according national guidelines without stem cells serves as comparator.

Diabetic foot patients with chronic limb ischemia and without the option for surgical or interventional revascularization were recruited and randomized to the transplant groups or the control group within this clinical trial. To measure the therapeutic effects of the various treatment arms patients were evaluated for (ankle brachial index (ABI), transcutaneous oxygen partial pressure (TcPO2), and reactive hyperemia (Blood Oxygen Level Dependent [BOLD]). Patients also underwent imaging with angiographic methods.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus Type 1 or 2
* Peripheral occlusive arterial disease stage III or IV (Fontaine) with chronical ischemia, chronic foot ulcer, degree of severity <5 (Wagner), older than 6 weeks, without acute wound infection
* Ulcer size 1 - 30cm2, in case of osteomyelitis only one bone should be affected no trend towards healing in the ulcer after one week of standard treatment
* Angiopathic or angioneuropathic diabetic foot syndrome with no possible option of operative or interventional revascularisation
* Age 18 - 80 years
* Declaration of patient consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The patient is alive, the patient has not undergone any major amputation, complete primary wound healing has been achieved, no ipsilateral relapse has occurred | 12 months

SECONDARY OUTCOMES:
Rate major amputations Rate of patients with complete ulcer healing Rate of treatment related complications Improvement of ankle brachial index (ABI) Improvement of transcutaneous oxygen partial pressure (TcPO2) Improvement of local perfusion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Diethelm Tschoepe, Prof Dr Dr, Principal Investigator — Herz- und Diabeteszentrum NRW
Locations (1):
- Herz- und Diabeteszentrum Nordrhein Westfalen, Bad Oeynhausen, Germany

REFERENCES:
- [Derived] Kirana S, Stratmann B, Prante C, Prohaska W, Koerperich H, Lammers D, Gastens MH, Quast T, Negrean M, Stirban OA, Nandrean SG, Gotting C, Minartz P, Kleesiek K, Tschoepe D. Autologous stem cell therapy in the treatment of limb ischaemia induced chronic tissue ulcers of diabetic foot patients. Int J Clin Pract. 2012 Apr;66(4):384-93. doi: 10.1111/j.1742-1241.2011.02886.x. Epub 2012 Jan 27. PMID 22284892